CLINICAL TRIAL: NCT01711086
Title: Double Blind Placebo Controlled Trial Checking the Safety and Efficacy of the Inspiromatic Inhaler in Comparison to the Aerolizer Inhaler When Delivering Formoterol
Brief Title: Safety and Efficacy of the Inspiromatic Inhaler in Comparison to the Aerolizer Inhaler When Delivering Formoterol
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guy Steuer (Other)
Collaborators: Schneider Children's Medical Center, Israel (Other); Inspiromedical Inc (Unknown)
Responsible Party: Sponsor-Investigator, Guy Steuer, Guy Steuer, M.D., Rabin Medical Center
Organization: Rabin Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0401-11-RMC
Record Dates: First submitted 2012-09-22; First posted 2012-10-22 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Asthma
Keywords: asthma; dry powder inhaler
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inspiromatic followed by Aerolizer (Active Comparator): volunteers will perform lung function pre and post Formoterol (a bronchodilator) inhalation. They will use either the Inspiromatic dry powder inhalers the delivery device. 3-60 days later participants will receive the same drug through the Aerolizer dry powder inhaler.
  Interventions: Device: Inspiromatic followed by Aerolizer
- Aerolizer followed by Inspiromatic (Active Comparator): volunteers will perform lung function pre and post Formoterol (a bronchodilator) inhalation. They will use either the Aerolizer dry powder inhalers the delivery device. 3-60 days later participants will receive the same drug through the Inspiromatic dry powder inhaler.
  Interventions: Device: Aerolizer Followed by Inspiromatic

INTERVENTIONS:
Device: Aerolizer Followed by Inspiromatic — Participants will receive Formoterol (Foradil) 12mcg via the Foradil Aerolizer inhaler while performing lung function as part of the and not differ from other routine follow-up
  Other Names: Foradil Inhaler
  Arms: Aerolizer followed by Inspiromatic
Device: Inspiromatic followed by Aerolizer — Participants will receive Formoterol (Foradil) 12mcg via the Inspiromatic dry powder inhaler while performing lung function instead of getting it via the Foradil Aerolizer
  Other Names: Inspiromatic dry powder experimental inhaler
  Arms: Inspiromatic followed by Aerolizer

SUMMARY:
Double-blind study, randomized, controlled, and crossover. Study recruited 30 volunteers with stable asthma aged 8-18 years. Participants will perform lung function as part of the routine follow-up then will receive a Foradil 12mcg either with an Aerolizer (a standard dry powder inhaler) or with the Inspiromatic (an active, breath synchronized innovative inhaler). 3-60 days later participants will receive the same drug through the other inhaler.

Pre and post treatment (15 min, 30 min, 60 min) Lung function results, drug levels in the blood, vital signs and side effects will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Children 8-18 years with Asthma
* 50<FEV1<80
* Can perform Spirometry

Exclusion Criteria:

* Poor cooperation
* Pregnancy
* Milk Allergy
* Other lung disease
* Prior familiarity with Aerolizer

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-10; Primary Completion 2012-11 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
FEV1 | We will measure FEV1 post treatment (15 min, 30 min, 60 min)
  Change in FEV1 from base line

SECONDARY OUTCOMES:
Vital signs | Pre treatment and than 15 minutes post treatment
  Change in heart rate, blood pressure

OTHER OUTCOMES:
Systemic absorption | 0 and 15 minutes post inhaltion
  K concentration, Glucose levels and drug level

CONTACTS AND LOCATIONS:
Overall Officials: Guy Steuer, M.D., Principal Investigator — Schneider Children Hospital
Locations (1):
- Schneider Children Hospital, Petah Tikva, Israel